CLINICAL TRIAL: NCT03667560
Title: Randomized and Blinded Clinical Evaluation of Dermacell Without Basement Membrane in Breast Reconstruction.
Brief Title: Dermacell ADM Without Basement Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20295
Record Dates: First submitted 2018-04-06; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: Mastectomy; Breast Reconstruction; Acellular dermal matrix
MeSH Terms: conditions — Breast Neoplasms | interventions — FlexHD

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dermacell ADM without basement membrane (Experimental): Dermacell ADM without a basement membrane
  Interventions: Procedure: Dermacell ADM without basement membrane
- FlexHD (Active Comparator): FDA-approved FlexHD Pliable
  Interventions: Procedure: FlexHD

INTERVENTIONS:
Procedure: Dermacell ADM without basement membrane — Patient will be implanted with Dermacell ADM.
  Arms: Dermacell ADM without basement membrane
Procedure: FlexHD — Patient will be implanted with FlexHD.
  Arms: FlexHD

SUMMARY:
DermACELL acellular dermal matrix (D-ADM) is the trade name of LifeNet Health's acellular dermal matrix (ADM). LifeNet Health will remove the basement membrane from the D-ADM and this product will be compared to FlexHD® Pliable, which does not include a basement membrane in order to demonstrate that D-ADM without a basement membrane is not inferior to FlexHD in the frequency of significant side effects that result from breast implants. This is a post market trial that is comparing two ADM products with a known safety profile. The D-ADM without a basement membrane is being prepared specifically for this UVA evaluation. Removal of the basement membrane by the manufacturer is considered minimal manipulation. D-ADM without a basement membrane will be considered a human cell, tissue, and cellular and tissue-based product (HCT/P) and is eligible for marketing immediately within the US, if desired by LifeNet Health (LNH). Additionally, the applications of the products are indicated. Therefore, the trial is not in support of an Investigational Device Exemption (IDE).

Prior to surgery, the registered subject will be randomized to receive the D-ADM without the basement membrane or the comparator, FlexHD Pliable. The surgeon and the patient will be blinded to the product group. The patient will receive the ADM at the time of placement of the tissue expander. After a period of tissue expansion, the patient will have the expander-implant exchange. During this surgery, there will be 3 punch biopsies taken in 3 different locations: native breast tissue, center of the ADM, and the border of the ADM and subject's breast tissue. These specimens will be analyzed to estimate differences in immunologic and inflammatory response for each ADM product.

The patient will follow up with the surgeon at 1-3 weeks, 3 months, 6 months, 9 months, and 12 months post implant exchange. At these visits, the surgeon will assess for any adverse events and this information will be collected for research purposes. The patient will be asked to complete the reconstruction module of the Breast-Q at the baseline visit and 6 and 12 months to assess quality of life and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer
* Candidate for and decide to undergo implant-based reconstruction
* Willing and able to provided written informed consent and comply with the study protocol.

Exclusion Criteria:

* Women planning to undergo radiation treatment or whose tumor characteristics of the mastectomy specimen dictate that post-op radiation will be required.
* Women planning to undergo adjuvant chemotherapy.
* Women who have had prior breast cancer treated with breast conservation therapy requiring radiation for the same breast being treated will be excluded.
* Known sensitivity to either of the following antibiotics: lincomycin, gentamicin, polymyxin B, or vancomycin.
* Women who have the presence of any condition that in the opinion of the investigator places the participant at undue risk or potentially jepordizes the quality of data to be generated.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Seroma Formation | 12 months
  Determine severity of seroma formation with each arm by observing drainage output and if seroma requires significant surgical intervention.

SECONDARY OUTCOMES:
Capsular Contracture | 12 months
  Estimate the degree of capsular contracture in participants in each study arm by using the Baker Scale.
  Grade I-The breast is soft and appears natural in size and shape. Grade II- The breast is slightly firm but appears normal Grade III- The breast is firm and appears abnormal Grade IV- the breast is hard, painful to the touch, and appears abnormal
Red breast syndrome | 12 months
  Estimate the frequency of red breast syndrome among participants on each arm
QOL | 12 months
  Determine patient's quality of life and satisfaction with the reconstruction process. Assessment will be done with the standardized Breast-Q Reconstruction Module.
Infection | 12 months
  Estimate the frequency and degree of infection among patients on each study arm. Infections will be identified by the surgeon and determined to be major or minor. In addition to this, the need for IV s. oral antibiotics and/or further surgery will be used as a measure of degree of infection.
Histological Assessment | Day 1
  Estimate the differences in immunologic and inflammatory responses on each study arm by histological assessment of the capsular and ADM biopsies, including quantity of inflammatory cells, macrophages, and migration/differentiation of myelofibroblasts.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No